CLINICAL TRIAL: NCT06285331
Title: the Impact of Manual or Mechanical Ways to Perform Passive Leg Raising on the Accuracy of Evaluation of Fluid Responsiveness
Brief Title: the Impact of Manual or Mechanical Ways to Perform PLR on the Accuracy of Evaluation of Fluid Responsiveness
Acronym: PLR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Zhongda Hospital, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023ZDSYLL483-P01
Record Dates: First submitted 2024-01-09; First posted 2024-02-29 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Circulatory Failure
Keywords: Fluid Responsiveness; Passive Leg Raising
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Bed (Active Comparator): PLR will be performed by adjusting the automatic bed the patients stay on.
  Interventions: Device: Automatic Bed
- Manual (Placebo Comparator): PLR will be performed by the investigators by their hands.
  Interventions: Device: Manual

INTERVENTIONS:
Device: Automatic Bed — The automatic bed is controlled by a screen and allows clinicians to perform passive leg raising on patients without touching them physically.
  Arms: Automatic Bed
Device: Manual — The clinicians will perform passive leg raising on patients by touching their legs physically.
  Arms: Manual

SUMMARY:
Our goal was to study the impact of different ways to perform passive leg raising (PLR) on the accuracy of evaluation of fluid responsiveness.

DETAILED DESCRIPTION:
Patients who have shock of all kinds of reasons usually need to be transferred to the Intensive Care Unit(ICU) for monitoring and treatment due to unstable vital signs and high fatal risks. The cardiac function of these patients requires special attention. Fluid responsiveness is a comprehensive reflection of preload and cardiac function, which provides guidance on how to conduct fluid replacement therapy. When patients have fluid responsiveness, it means that after fluid resuscitation therapy, the patients' cardiac output will increase and tissue perfusion will improve, bringing benefits to patients themselves. Therefore, it is of vital significance to evaluate the presence of fluid responsiveness in patients before fluid therapy in clinical practice. Passive leg raising(PLR) is a commonly used method in clinical practice to evaluate patients' fluid responsiveness. But its accuracy is affected by the way the leg lifting is performed.

This project is aimed to explore the impact of different ways to perform passive leg raising on the accuracy of evaluation of fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients who have signs of tissue hypo-perfusion (increasing lactate levels, in need of vasopressor agents to maintain blood pressure, oliguria, and weak consciousness), and need to evaluate their fluid responsiveness; (2) patients who have received Pulse indicator Continuous Cardiac Output (PiCCO) monitoring ; (3) patients who are transferred into the intensive care department.

Exclusion Criteria:

* (1) Age < 18 years old, or > 75 years old (2) pregnancy or lactation; (3) refusal to sign the informed consent form for enrollment; (4) patients who are clearly unable to perform passive leg raising (PLR) (intra-abdominal pressure ≥16cmH2O, high risk of lower limb venous thrombosis, intracranial hypertension, and recent undergone abdominal or pelvic surgery); (5) patients with the contraindications of fluid resuscitation therapy ( pulmonary edema, intracranial hypertension and so on); (6) patients clinical doctors assessed as unsuitable for PLR.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of fluid responsiveness evaluation | Immediately after procedure
  It is the results of accuracy of evaluation of patients' fluid responsiveness by performing PLR by different ways. The accuracy is evaluated by comparing the results of PLR and fluid challenge test. The cardio output of patients is obtained by Pulse indicator Continuous Cardiac Output (PiCCO). The results of PLR are considered accurate if the results of the patient's volume responsiveness measured by different methods of PLR are consistent with the results obtained by the fluid challenge test.

SECONDARY OUTCOMES:
Mortality | 90days
  The mortality of patients within 90 days after PLR was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China